CLINICAL TRIAL: NCT03600493
Title: Comparison Between Dexmedetomidine and Lidocaine as an Adjuvant to General Anesthesia in Patients Undergoing Major Abdominal Surgeries
Brief Title: Adjuvant to General Anesthesia in Patients Undergoing Major Abdominal Surgeries
Acronym: Adjuvant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mohamed A Elsadany, MD, Principal Investigator, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3399
Record Dates: First submitted 2018-07-02; First posted 2018-07-26 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Stress Related Disorder
MeSH Terms: interventions — Dexmedetomidine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexemetomidine (Active Comparator): Dexmedetomidine 1 mcg/kg over 10 min followed by 0.4 mcg/kg/hr. till the start of wound closure.
  Interventions: Drug: Dexmedetomidine
- Lidocaine (Active Comparator): Lidocaine prepared in a syringe with the same volume of Dexmedetomidine to assure blinding given as 1mg/kg over 10 min followed by 1mg/kg/hr till the start of wound closure.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 1 mcg/kg over 10 min followed by 0.4 mcg/kg/hr. till the start of wound closure.
  Other Names: Selective Alpha 2 agonist
  Arms: Dexemetomidine
Drug: Lidocaine — Lidocaine given as 1mg/kg over 10 min followed by 1mg/kg/hr till the start of wound closure.
  Other Names: Lignocaine
  Arms: Lidocaine

SUMMARY:
assessing the effect of perioperative infusion of Dexmedetomidine versus Lidocaine on neuro endocrine stress response to surgery and anesthesia

DETAILED DESCRIPTION:
Methodolgy

During the preoperative visit, the techniques will be explained to patients including benefits and complications.

1) Pre-operative assessment:

A) Medical history:

1. Medical disorders as hypertension, diabetes, heart, chest, liver or kidney diseases.
2. Past history of operations, hospitalization or blood transfusion.
3. Past anesthetic history with impact on previous airway problems during previous surgeries, hypersensitivity to anesthetic medications, any previous post-operative complications that could be attributed to anesthesia.
4. Family history for specific anesthetic problems like malignant hyperthermia.

B) Physical examination:

1. General examination, & vital signs (heart rate, blood pressure, respiratory rate and temperature) in bed the night before operation
2. Heart, chest and abdominal examinations

C) Anesthetic assessment:

1. Examination of the limbs for prediction of difficult cannulation.
2. Airway assessment including:

   1. Thyromental distance
   2. Mallampatti score
   3. Neck and tempro-mandibular joint mobility
   4. Assessing the absence of deformities in the mandible, face, tongue, palate, teeth and neck that may interfere with airway management

D) Laboratory investigations:

* Complete blood count
* Prothrombin time and partial tissue thromboplastic time
* Kidney function test (s, creatinine & urea), Liver function test (ALT, AST, albumin and bilirubin) & Random blood sugar.
* Serum Cortisol and IL6 level before starting drug infusion.

  2) Demographic data: The patient's age, sex, ASA status, and duration of surgery will be recorded.

  3) Technique:
  1. Patients will be fasting for 6 - 8 hours.
  2. All patients will receive oral midazolam (7.5 mg), and oral ranitidine (150mg) administered 90 min before arrival in the operating room with a sip of water.
  3. All patients will receive a pre-induction normal saline 10 ml/kg body weight over 10-15 minutes. Subsequently, intravenous fluid administration will be done according to the need of each patient.
  4. All operations will start between 08.30 am and 09.30 am, to minimize variations in cortisol level.
  5. All patients will receive the drug of study 10 min before induction of anesthesia till the start of wound closure in the form of:

     Group (D) Dexmedetomidine 1 mcg/kg over 10 min followed by 0.4 mcg/kg/hr. till the end of wound closure.

     Group (L) Lidocaine prepared in a syringe with the same volume of Dexmedetomidine to assure blinding given as 1mg/kg over 10 min followed by 1mg/kg/hr.
  6. Doses will be calculated, diluted in 50 ml of normal saline and given intravenously by a syringe pump over 10 minutes initially and then over 1hr till the start of wound closure.
  7. All drugs of the study will be prepared by an independent anesthesiologist who will not share in the study and then selected and given by another one blinded for the content of each syringe.
  8. Airway devices, anesthesia machine, ventilator, flowmeters and monitors will be checked promptly.
  9. Another wide-bore I.V cannula will be inserted in case of blood transfusion.
  10. Monitoring equipment's (Datex-Ohmeda™) will be attached to the patient including 3-leads ECG, non-invasive arterial blood pressure, pulse oximetery and capnograph after tracheal intubation.
  11. The depth of anesthesia will be monitored with Entropy device. The Entropy electrodes will be placed on the forehead and on the lateral angle of orbit and connected to (Datex-Ohmeda™) by a special. The target Entropy range will be 40-60 for surgical anesthesia.
  12. Induction of anesthesia will be performed by Propofol 2 mg/kg followed by cis-atracurium 0.15 mg/kg and fentanyl 1 mcg/kg given intravenously after pre-oxygenation with 100% oxygen for at least 3 minutes.
  13. Patients will be manually ventilated with 100% oxygen till intubation after 2 min and with Entropy value of 60 to 40 by Macintosh laryngoscope and appropriate size endotracheal tube.
  14. Maintenance of anesthesia will be carried out by isoflurane varying its end tidal concentration to keep Entropy in the range of 55 to 40 with Air:Oxygen mixture 0.3 fraction of oxygen and flow rate of 2 liter in completely closed circuit.
  15. Cis-atracurium 0.03 mg/kg guided by neuromuscular monitor Train of Four (TOF) will be used for muscle relaxation.
  16. Hemodynamics (mean arterial blood pressure and heart rate) will be maintained within 25 % of baseline measures.
  17. Any increase of MAP or HR more than 25% of baseline measures on two consecutive readings within 2-3 min will be managed by I.V bolus of fentanyl 0.5 mcg/kg and any decrease of MAP or HR less than 25 % on two consecutive readings within 2-3 min will be managed by I.V bolus of ephedrine 5 mg or atropine 0.5 mg respectively.
  18. The infusion of study medication will be discontinued if the hypotension persisted > 5 min after these interventions upon return of the MAP or HR to within 25% of the baseline value, the study medication infusion will be resumed at 50% of the initial infusion rate and then gradually increased to the initial infusion rate.
  19. The infusion of study medication will be discontinued at the start of wound closure. Upon completion of wound closure, isoflurane will be discontinued and the inspired oxygen flow rate will be increased to 5 L/min and residual neuromuscular block will be reversed with neostigmine, 0.05 mg/kg IV, and atropine 0.25 mg/kg, IV. The trachea will be extubated when the patient is fully awake. Transfer to the recovery room will be done when the patient scored 7 and above using the modified Aldrete scoring system.
  20. On emergence from anesthesia and immediately in post anesthesia care unit, analgesic regimen, consisting of intravenous patient-controlled morphine analgesia (bolus 1mg, 10-min lockout, maximum dose 5 mg / h), will be used in all groups.
  21. The whole technique and anesthetic procedures will be performed by the same anesthesiologist to avoid as much as possible the inter-individual skill variations.

ELIGIBILITY:
Inclusion Criteria:

* Both gender.
* Consent from patients about technique and nature of the study.
* Patients are ASA I (American Society of Anesthesiology physical status Grade I) = (normal healthy patients) or ASA II (American Society of Anesthesiologists physical status Grade II).
* Patients scheduled for major abdominal surgery.

Exclusion Criteria:

1. Pre-operative regular medication with opioids and benzodiazepines, alcohol abuse, known sleep disturbance, known endocrine disease
2. Known allergy to Dexmedetomidine or Lidocaine.
3. History of endocrine disorders.
4. Heart block greater than first degree.
5. Medication known to affect the sympathetic response or hormonal secretion.
6. Smokers.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Interleukin 6 (IL6) | Serum Interleukin 6 will be measured at baseline and then 2 hours after induction of surgery and then 6 hours postoperative
  Serum Interleukin 6 will be measured in picogram/Milliliter

SECONDARY OUTCOMES:
Change in Serum Cortisol | Serum Cortisol will be measured as baseline and then 2 hours after induction of surgery and then 6 hours postoperative
  Measurement of Serum Cortisol levels in microgram/deciliter
Changes in Mean Arterial Blood Pressure (MABP) | Baseline MABP, immediately before induction and 1, 2, 3 and 5 min after intubation, then immediately before extubation, 1, 2, 3 and 5 min after extubation
  MABP changes in mmHg with intubation, extubation and throughout surgery
Changes in Heart Rate (HR) | Baseline HR, immediately before induction and 1, 2, 3 and 5 min after intubation, then immediately before extubation, 1, 2, 3 and 5 min after extubation
  HR changes with intubation, extubation and throughout surgery
Morphine consumption | Morphine consumption during first 24 hours postoperatively
  Total postoperative morphine consumption in mg during first 24 hours
Ephedrine | During intraoperative period
  Total Ephedrine dose in mg used intraoperative for treatment of hypotension
Atropine consumption using questionnaire | During intraoperative period
  Total Atropine dose in mg used intraoperative for treatment of bradycardia
Visual analogue scale VAS | VAS (visual analogue scale) at 1, 2, 4, 8, 12 and 24 hours postoperatively.
  Pain scale measurement for postoperative assessment of pain consisting from 0 to 10 representing 0 as no pain and 10 as the most imaginable pain treating the patient if VAS > 3

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Elsadany, MD, Principal Investigator — Anesthesia and Intesive Care department, Faculty of Medicine, Suez Canal University